CLINICAL TRIAL: NCT01157208
Title: Dietary Interventions for Chronic Daily Headache (CDH): A Feasibility Study,
Brief Title: Nutrition for Chronic Daily Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Mayday Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-0600
Record Dates: First submitted 2010-05-28; First posted 2010-07-05 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2012-11

CONDITIONS: Chronic Daily Headache
Keywords: chronic pain; headache; nutrition; inflammation; complementary medicine
MeSH Terms: conditions — Headache Disorders; Chronic Pain; Headache; Inflammation | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet A (Experimental): This diet is high in omega-3 fatty acids, low in trans fatty acids, and low in omega-6 fatty acids. Subjects are encouraged to eat fatty fish daily (e.g., salmon), to limit vegetable oil intake, and to eat fruits, vegetables and whole grains. Specifically formulated and other provided foods for this group will include salmon-salad sandwiches, hummus with olive oil, other bean dips and bean dishes, frozen and canned fish, and blueberry-flax muffins.
  Interventions: Other: Diet A
- Diet B (Experimental): This diet is low in trans fatty acids and low in omega-6 fatty acids. Subjects are encouraged to to limit vegetable oil intake, to replace meats and eggs with beans and lean fish/shellfish, and to eat fruits, vegetables and whole grains. Specifically formulated and other provided foods for this group will include hummus with olive oil, other bean dips and bean dishes, lean fish and shellfish,and blueberry muffins.
  Interventions: Other: Diet B

INTERVENTIONS:
Other: Diet A — Subjects receive dietary counseling, food for two meals and two snacks daily, and access to a website with recipes, approved food lists, and dining out guides for a 12-week intervention.
  Other Names: nutrition
  Arms: Diet A
Other: Diet B — Over a 12-week intervention, subjects receive dietary counseling, food for two meals and two snacks daily, and access to a website with recipes, approved food lists, and dining out guides.
  Other Names: nutrition
  Arms: Diet B

SUMMARY:
The purpose of this study is: 1) To assess the feasibility of implementing a clinical trial comparing two potentially analgesic dietary interventions in patients with chronic daily headache (CDH) and 2)To assess the preliminary efficacy of the dietary interventions on headache frequency and severity and 3) to assess the impact of the diet on the percentage of omega-6 highly unsaturated fatty acids (HUFA) in total HUFA in whole blood.

During a 6-week baseline phase, eligible individuals with CDH will complete web-based daily diaries, self-report questionnaires, and nutrient intake assessments. Before randomization to one of the two intervention groups, blood will be collected to measure baseline nutritional biomarkers. Targeted dietary advice will be administered and foods will be provided throughout the 12-week intervention phase. Samples for biomarkers will be collected every 4 weeks during the intervention. Participants will continue recording headache characteristics with a daily headache diary. At the conclusion of the intervention, participants will provide complete follow-up assessments and blood for nutritional biomarker measurement.

DETAILED DESCRIPTION:
CDH is characterized by structural and functional immune and nervous system derangements. Specifically, disturbed regulation of the following critically important biochemical processes has been demonstrated: 1) inflammation; 2) neuronal membrane excitability; and 3) monoamine neurotransmitter signaling. Accordingly, major classes of medications used for chronic pain (anti-inflammatories, anticonvulsants, and antidepressants) target these processes.

Foods consist of combinations of nutrient molecules that are incorporated into human tissues, and enter into and regulate highly leveraged human biochemical pathways. By altering the structure and function of the nervous system and immune system, and regulating biochemical processes believed to play causal roles in the development and maintenance of chronic pain, dietary choices may play a critical role in the initiation and/or perpetuation of CDH.

Multifaceted, targeted dietary manipulation, directed towards correcting underlying biochemical derangements, represents a novel therapeutic approach to the management of chronic pain. Improved understanding of the relationships between dietary selections and chronic pain promises to benefit the estimated 10 million Americans with CDH and possibly an even larger population with chronic pain from any origin. For a more detailed description, please refer to the complete rationale and literature review accompanying grant application.

Major research questions for this proposal include:

A. Is it possible to implement a controlled dietary trial comparing two analgesic dietary interventions for subject with CDH? and B. What are the preliminary estimates of impact of targeted analgesic dietary interventions on headache frequency compared with one another and the baseline headache frequency in patients for CDH? C. What is the rate and extent of change in %n6 in HUFA with two targeted interventions? There is also an exploratory portion of the study to gather more information about the potential relationship between nutrient and pain to inform intended future trials. The study is needed to assess the potential utility of a dietary approach for chronic pain, which may have major public health implications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* either gender
* meeting the 2004 International Classification of Headache Disorders (ICHD - II) criteria for the following forms of CDH (15 or more headache days per month and a headache history of more than two years with chronic migraine, transformed episodic migraine into CDH, chronic tension-type headache and new persistent daily headache)
* under the care of a neurologist
* willing and able to document headache characteristics and use of medications, as well as complete the assessment instruments
* able to come in for 3 dietitian-administered dietary counseling sessions over 12 weeks
* able to speak and understand English

Exclusion Criteria:

* analgesic rebound headache
* hemicrania continua
* drug-induced headache
* post-traumatic headache
* significant, symptomatic uncontrolled psychosis
* undergoing current treatment for a major medical illness such as malignancy, autoimmune or immune deficiency disorder
* pregnancy
* clotting disorders
* history of cranial or neck surgery within two years
* vasculitis
* chronic subdural hematoma
* history of meningitis
* history of subarachnoid or intracerebral hemorrhage
* history of eating disorder
* regular use of supplemental omega-3 fatty acids or gamma-linolenic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Headache Impact Test | Pre-intervention and post-intervention
  Headache-related quality-of-life measure

SECONDARY OUTCOMES:
Omega-3 and omega-6 fatty acids in RBCs and plasma | pre-intervention and at 4 and 8 weeks, and at the conclusion of the intervention.
  Highly-unsaturated fatty acids are measured in plasma and red blood cells before the intervention, during the intervention at 4 and 8 weeks, and at the conclusion of the intervention at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: John Douglas Mann, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data has been shared with NIH.

REFERENCES:
- [Result] Ramsden CE, Faurot KR, Zamora D, Palsson OS, MacIntosh BA, Gaylord S, Taha AY, Rapoport SI, Hibbeln JR, Davis JM, Mann JD. Targeted alterations in dietary n-3 and n-6 fatty acids improve life functioning and reduce psychological distress among patients with chronic headache: a secondary analysis of a randomized trial. Pain. 2015 Apr;156(4):587-596. doi: 10.1097/01.j.pain.0000460348.84965.47. PMID 25790451
- [Result] Ramsden CE, Faurot KR, Zamora D, Suchindran CM, MacIntosh BA, Gaylord S, Ringel A, Hibbeln JR, Feldstein AE, Mori TA, Barden A, Lynch C, Coble R, Mas E, Palsson O, Barrow DA, Mann DJ. Targeted alteration of dietary n-3 and n-6 fatty acids for the treatment of chronic headaches: a randomized trial. Pain. 2013 Nov;154(11):2441-2451. doi: 10.1016/j.pain.2013.07.028. Epub 2013 Jul 22. PMID 23886520
- [Derived] Ramsden CE, Zamora D, Makriyannis A, Wood JT, Mann JD, Faurot KR, MacIntosh BA, Majchrzak-Hong SF, Gross JR, Courville AB, Davis JM, Hibbeln JR. Diet-induced changes in n-3- and n-6-derived endocannabinoids and reductions in headache pain and psychological distress. J Pain. 2015 Aug;16(8):707-16. doi: 10.1016/j.jpain.2015.04.007. Epub 2015 May 7. PMID 25958314
- [Derived] Ramsden CE, Mann JD, Faurot KR, Lynch C, Imam ST, MacIntosh BA, Hibbeln JR, Loewke J, Smith S, Coble R, Suchindran C, Gaylord SA. Low omega-6 vs. low omega-6 plus high omega-3 dietary intervention for chronic daily headache: protocol for a randomized clinical trial. Trials. 2011 Apr 15;12:97. doi: 10.1186/1745-6215-12-97. PMID 21496264